CLINICAL TRIAL: NCT02812043
Title: Comparison of the Efficacy and Safety Between Long-pulsed Nd:YAG, Amorolfine and Combination of Long-pulsed Nd:YAG and Amorolfine in Treating Non-dermatophyte and Mixed-infection Onychomycosis
Brief Title: Comparison Between Long-pulsed Nd:YAG, Amorolfine and Combination Treatment in Treating Non-dermatophyte Onychomycosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 391/2558(EC1)
Record Dates: First submitted 2015-10-13; First posted 2016-06-23 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Non-dermatophyte Onychomycosis
Keywords: onychomycosis; amorolfine; long-pulsed Nd:YAG; fungal infection
MeSH Terms: conditions — Onychomycosis; Mycoses | interventions — amorolfine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Amorolfine (Experimental): This group of patients will receive only amorolfine nail lacquer to apply on the affected nail and the KOH examination and fungal culture will be performed every month
  Interventions: Drug: Amorolfine
- Long-pulsed Nd:YAG (Experimental): This group of patients will receive only the long-pulsed Nd:YAG (Cynergy®, 5 Carlisle Road Westford, MA USA) fluence 35-45 J/Cm2, spot size 4mm for 2 passes each visit with 4-week intervals and the KOH examination and fungal culture will be performed every month
  Interventions: Device: 1,064nm Long-pulsed Nd:YAG
- Amorolfine+Long-pulsed Nd:YAG (Experimental): This group of patients will receive both amorolfine nail lacquer and the long-pulsed Nd:YAG laser treatment each visit with 4-week intervals and the KOH examination and fungal culture will be performed every month
  Interventions: Device: 1,064nm Long-pulsed Nd:YAG; Drug: Amorolfine

INTERVENTIONS:
Device: 1,064nm Long-pulsed Nd:YAG — Long-pulsed 1,064nm will be used for the treatment of onychomycosis which wll use 35-45 J/cm2 spot size 4, frequency 1 Hz for 2 passes on the infected nails
  Other Names: Dualis SP; Fotona, Lujbljana
  Arms: Amorolfine+Long-pulsed Nd:YAG; Long-pulsed Nd:YAG
Drug: Amorolfine — Amorolfine nail lacquer will be applied by the patient once a week on the infected nails
  Arms: Amorolfine; Amorolfine+Long-pulsed Nd:YAG

SUMMARY:
This study aims to compare the efficacy and safety of amorolfine, long-pulsed Nd:YAG laser and the combination between amorolfine and long-pulsed Nd:YAG in treating the non-dermatophyte and mixed-infection onychomycosis.

DETAILED DESCRIPTION:
Onychomycosis is the most common cause of nail deformities resulting with more than 50% of the patients with abnormal nails. From the institution of dermatology of Thailand, it confirmed that 1.7% of Thai population have onychomycosis. Most of the patients aged between 40-60 years old with female predominated. The common cause of onychomycosis worldwide is dermatophyte group, found in more than 50% of the patients. However, in Thailand, the study showed that 51.6% of patients with onychomycosis were infected by non-dermatophyte group especially Neoscytalidium spp.

The goal standard treatment for onychomycosis was oral anti-fungal drugs such as Fluconazole, Itraconazole and Terbinafine. But many patients were limited to the oral medications due to drug interaction between other CYP P2C9 inhibition such as statins, causing the risk of rhabdomyolysis and hepatotoxicity. Even though these medications are effective against dermatophytes. The non-dermatophytes which were the leading pathogens for onychomycosis in Thailand tends to be resistant to the oral medications. Therefore topical and other modalities have become an important role for treating those non-dermatophytes onychomycosis such as topical anti-fungals, topical urea cream and laser treatment. So far, no standard treatment has been made in order to treat the non-dermatophyte onychomycosis causing problems to both patients and physicians in Thailand.

Amorolfine is a morpholine derivative used in topical anti-fungal that inhibits the biosynthesis of the fungal cell membrane and showed fungicidal activities. From the previous study, amorolfine is an effective topical treatment against non-dermatophyte onychomycosis with 52-55% mycological cure rate and the clinical cure rate varied from 12.7%-54% depending on the studies. The side effects were minimal and the application was simple to use. So amorolfine is used as a first line treatment for non-dermatophyte onychomycosis in our practice. However, with the long treatment (from 6 months up to 1 year) and the low mycological cure rate newer modality had been studied to deal with this problematic pathogens.

Long-pulsed Nd:YAG laser had been used to treat onychomycosis with a promising result. In 2013, Kostas Kalokasidis used long-pulsed Nd:YAG for the onychomycosis and showed a 94.5% mycological cure rate with no relapse of the disease within 3 months. Later on, Rungsima Wanitphakdeedecha M.D. tried the long-pulsed Nd:YAG to treat onychomycosis and found the significant result that long-pulsed Nd:YAG can cure up to 95.42% onychomycosis from non-dermatophyte group. But the protocol was performed the laser treatment every 2 weeks for 1 month which made it difficult for the patient to come to the hospital, moreover the duration to treat onychomycosis might needed to be longer.

So the investigators came up with this study to compare the efficacy of long-pulsed Nd:YAG with 4-week intervals to the amorolfine and the combination of both Nd:YAG and amorolfine to see the mycological result and also the clinical improvement.

The treatment and KOH examination and fungal culture will be performed every month for 4 months, and then the follow up will be at 6 months after the first treatment

ELIGIBILITY:
Inclusion Criteria:

1. The patients aged more than 18 years old.
2. The patients were diagnosed with non-dermatophytes or mixed-infection onychomycosis from both KOH examination and fungal cultured.
3. The patients did not have any prior anti-fungal treatment within 6 months
4. The patients did not receive any vasodilator drugs or isotretinoin within 6 months
5. The patients who are willing to participate, and accept the methods and risk

Exclusion Criteria:

1. The patients who suffered other medical dermatologic condition associated with onychomycosis such as psoriasis, paronychia etc.
2. The patients who took immunosuppressive drugs, or the immunocompromised host.
3. The patients who had severe vascular disease, such as severe DVT, or poor capillary refill time.
4. The patients who had onychomycosis which involved in nail matrix.
5. Pregnancy or lactation.
6. The patients who had problems communication or have difficulty travel to the faculty for the checkup.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Mycological cure rate in patients with onychomycosis after Amorolfine, long-pulsed Nd:YAG and the adjunct treatment | 6 months after treatment
  Mycological cure defined as negative Mycological culture

SECONDARY OUTCOMES:
Mycological cure rate in patients with onychomycosis after Amorolfine, long-pulsed Nd:YAG and the adjunct treatment | 1 month after treatment
  Mycological cure rate
Mycological cure rate in patients with onychomycosis after Amorolfine, long-pulsed Nd:YAG and the adjunct treatment | 2 months after treatment
  Mycological cure rate
Mycological cure rate in patients with onychomycosis after Amorolfine, long-pulsed Nd:YAG and the adjunct treatment | 3 months after treatment
  Mycological cure rate
number of participants who develop paronychia after Amorolfine, long-pulsed Nd:YAG and the adjunct treatment | 1 month after treatment
  number of participants
number of participants who develop paronychia after Amorolfine, long-pulsed Nd:YAG and the adjunct treatment | 2 months after treatment
  number of participants
number of participants who develop paronychia after Amorolfine, long-pulsed Nd:YAG and the adjunct treatment | 3 months after treatment
  number of participants
number of participants who develop paronychia after Amorolfine, long-pulsed Nd:YAG and the adjunct treatment | 6 months after treatment
  number of participants
pain score in participants who received long-pulsed Nd:YAG and the adjunct treatment | 1 month after treatment
  pain score
pain score in participants who received long-pulsed Nd:YAG and the adjunct treatment | 2 months after treatment
  pain score
pain score in participants who received long-pulsed Nd:YAG and the adjunct treatment | 3 months after treatment
  pain score
pain score in participants who received long-pulsed Nd:YAG and the adjunct treatment | 4 months after treatment
  pain score
Depth of nail involvement of onychomycosis after Amorolfine, long-pulsed Nd:YAG and the adjunct treatment | 1 month after treatment
  Depth of nail
Depth of nail involvement of onychomycosis after Amorolfine, long-pulsed Nd:YAG and the adjunct treatment | 2 months after treatment
  Depth of nail
Depth of nail involvement of onychomycosis after Amorolfine, long-pulsed Nd:YAG and the adjunct treatment | 3 months after treatment
  Depth of nail
Depth of nail involvement of onychomycosis after Amorolfine, long-pulsed Nd:YAG and the adjunct treatment | 6 months after treatment
  Depth of nail

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology Siriraj Hospital, Bangkoknoi, Bangkok, Thailand